CLINICAL TRIAL: NCT02689557
Title: VEINEX : Venous Investigations During Exercise
Acronym: VEINEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01440-47
Record Dates: First submitted 2016-02-11; First posted 2016-02-24 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- measures of the volumes (Other): Measures of the volumes of the lower limbs. A measure to rest, a measure of effort (walk) and a measure recovery. Intervention.
  Interventions: Other: plethysmography

INTERVENTIONS:
Other: plethysmography — Validate the measurement made by electroactive polymer sensors (plethysmography) during walking tests in venous insufficient subjects and healthy subjects by comparing the measurement made by the reference technique by mercury gauge.

SUMMARY:
Successfully develop and confirm with the Higher School of Electronics West Plethysmographic a multichannel recorder to perform measurements staggered volume of the lower limbs at rest, walking and recovery (6 storied measures on members lower).

DETAILED DESCRIPTION:
Validate the measurement made by EAP (Electroactive polymer) during walking tests in venous insufficient subjects and healthy subjects by comparing the measurement made by the reference technique by mercury gauge.

ELIGIBILITY:
Inclusion Criteria:

* present or not venous pathology

Exclusion Criteria:

* amputation of a lower limb
* heart failure
* Severe respiratory disease
* Unstable angina or myocardial infarction
* Parkinson's disease, hemiplegia and paraplegia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
plethysmographic record for volume measurement of lower limbs at rest, walking and recovery (6 measures stepped on the lower limbs) | Maximum 3 months
  plethysmographic record for volume measurement of lower limbs at rest, walking and recovery (6 measures stepped on the lower limbs)

CONTACTS AND LOCATIONS:
Overall Officials: ANTOINE BRUNEAU, MD, Principal Investigator — UH ANGERS
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No